CLINICAL TRIAL: NCT05966506
Title: A Culturally Adapted, Social Support-Based, Physical Activity Interventions for South Asian Indian Women in the United States: A Feasibility Study
Brief Title: A Culturally Adapted, Social Support-Based, Physical Activity Interventions for South Asian Indian Women in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nitha Mathew Joseph, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SN-23-0576; UL1TR003167-04 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Sedentary Behavior
Keywords: physical activity; social support
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health coaching (Experimental)
  Interventions: Behavioral: Dyad-based Zoom health coaching; Behavioral: Fitbit activity monitor; Other: Electronic newsletters

INTERVENTIONS:
Behavioral: Dyad-based Zoom health coaching — This will be delivered by a certified nurse coach, certified in holistic nursing who will provide 6 sessions of Zoom health coaching over 12 weeks to dyads, biweekly (weeks 1, 3, 5,7, 9 &11) for 45 minutes
Behavioral: Fitbit activity monitor — Participants will be instructed to use the Fitbit to monitor their partners' PA in addition to their own. All participants will be instructed to "friend" their health coach to enable real-time monitoring of PA to inform coaching zoom calls. The Fitbit will provide feedback on steps, active minutes, and calories burned. Participants will be asked to wear the device on most days and while they sleep.
Other: Electronic newsletters — Newsletters will be sent twice monthly during months 1-3 via email or text with an online link. Newsletters will be designed to share educational PA-related information from publicly available resources. Newsletters will also contain tips for overcoming barriers to PA ,finding time to exercise, low-cost ways to be active and being active with kids.Newsletters will also contain links to brief exercise routines that participants can do in their homes and information on low cost/free exercise classes in the community, which may help to overcome perceived access barriers

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of a peer-based dyadic social support health coaching physical activity (PA) intervention in inactive South Asian Indian (SAI) and to explore preliminary effects of the intervention on intermediate outcomes: self-reported and objective moderate-to-vigorous physical activity (MVPA), social support, and self-efficacy .

ELIGIBILITY:
Inclusion Criteria:

* inactive SAI (Physical activity (PA) <150 minutes/week)
* physically able to engage in moderate PA
* speak and read English; able to enroll with an eligible adult female partner who does not live in the same household
* willing to use the Fitbit app/device
* own a smartphone that is compatible with Fitbit software (up to 223.3 MB on iPhone or 165 MB on Android) 9)
* able and willing to send and receive text messages
* Blood pressure reading <160/100 mm Hg, or with medical clearance.

Exclusion Criteria:

* SAI women with a current/planned pregnancy
* cannot speak and read English
* those participating in a PA or weight loss program
* those diagnosed with a physical disability that interferes with their ability to be physically active.
* not living in Houston, Texas

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitha Mathew Joseph, PhD, RN, CNE, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty individuals (10 dyads) were enrolled in total: 10 participants, each enrolled with a study partner.
Period: Overall Study
Arm/Group | Health Coaching
Started | 20 (Twenty individuals (10 dyads) were enrolled in total: 10 participants, each enrolled with a study partner.)
Completed | 20 (Twenty individuals (10 dyads) were enrolled in total: 10 participants, each enrolled with a study partner.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes all twenty individuals enrolled (participants and their study partners).
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  South Asian Indian | 20
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 30.31 (5.36)
Education [Count of Participants; unit: Participants]
  Associates | 1
  Bachelors | 6
  Masters | 11
  Professional | 2
Annual Household Income [Count of Participants; unit: Participants]
  $50,000 to $79,999 | 1
  $80,000 to $99,999 | 2
  $100,000 or more | 17
Number of Participants Employed [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by the Percentage of Participants Enrolled in the Study
Time Frame: 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Number; unit: percentage of participants
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
percentage of participants | 100

2. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Complete the Study
Time Frame: 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
Participants | 20

3. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Complete All the Assessments
Description: Assessments include counseling calls ,use of Fitbit, receipt and review of newsletters
Time Frame: 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
Participants | 18

4. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Adhere to Treatment
Time Frame: 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
Participants | 18

5. Secondary Outcome: Physical Activity (PA) as Assessed by the Modified Godin Leisure-Time Exercise Questionnaire
Description: A modified version of the validated Leisure Score Index from the Godin Leisure-Time Exercise Questionnaire (GLTEQ) was used to assess episodes, intensity, and duration of PA during a typical 7-day period within the past month. The modified GLTEQ asked the participants to recall the amount of time spent in strenuous, moderate, and mild physical activity for each day over seven days. Time spent in moderate and strenuous physical activity was summed to calculate minutes of moderate-to-vigorous activity from the modified GLTEQ. Responses to the GLTEQ at each of the study assessments were converted to estimated weekly metabolic equivalent (METS). Responses on the LTEQ were converted into estimated weekly METS using a slightly modified version of the formula used by the developers of the GLTEQ: [(total METS = minutes of strenuous exercise / 15) × 9] + [(total minutes of moderate exercise / 15) × 5] + [(total minutes of light exercise / 15) × 3].
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: Weekly metabolic equivalent (METS)
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
Weekly metabolic equivalent (METS)
  Baseline | 23.85 (33.60)
  12 weeks | 53.37 (35.02)

6. Secondary Outcome: Physical Activity as Assessed by the Average Steps Per Day Measured Via Fitbit
Description: The average steps per day will be reported.
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
steps per day
  Baseline | 8,014 (2,705)
  12 weeks | 7,885 (4,091)

7. Secondary Outcome: Self-efficacy for Physical Activity as Assessed by the Self-efficacy for Physical Activity (SEPA) Scale
Description: The Self-efficacy for physical activity scale total score ranges from 5 to 25, a higher score indicating more confidence in one's ability to engage in physical activity
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale
  Baseline | 11.45 (4.25)
  12 Weeks | 12.95 (3.99)

8. Secondary Outcome: Physical Activity-related Social Support as Assessed by the Social Support for Physical Activity Survey (Study Partner Subscale)
Description: The Social Support for Physical Activity survey assess the level of support for exercising from both the individual (self) and their study partner. All participants completed both subscales: self-support subscale and study partner support subscale. Each subscale total score ranges from 13 to 104, with higher scores indicating greater social support. The study partner support subscale is reported.
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale
  Baseline | 16.45 (8.27)
  12 weeks | 31.75 (8.01)

9. Secondary Outcome: Physical Activity-related Social Support as Assessed by the Social Support for Physical Activity Survey (Self Support Subscale)
Description: The Social Support for Physical Activity survey assess the level of support for exercising from both the individual (self) and their study partner. All participants completed both subscales: self-support subscale and study partner support subscale. The survey consists of two subscales: self-support and study partner support. Each subscale total score ranges from 13 to 104, with higher scores indicating greater social support. The self support subscale is reported.
Time Frame: Baseline, 12 weeks
Population: Data was not collected from 1 individual in the health coaching arm at 12 weeks because the participant did not fill out that portion of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale
  Baseline | 14.3 (5.36)
  12 weeks: number analyzed (Participants) | 19
  12 weeks | 29 (8.23)

10. Secondary Outcome: Physical Activity Related Autonomy Support as Assessed by the Climate Questionnaire (Autonomy Support - Study Partner Subscale)
Description: The Climate questionnaire (autonomy support) asses the level of autonomy support provided by both the individual (self) and their study partner. All participants completed both subscales: self-support and study partner support. The study partner subscale is a 6 item questionnaire and each is scored from 1 (strongly disagree) to 7 (strongly agree). The sum of the 6 items were divided by 6, to generate a scale from 1 to 7, with higher scores indicating greater autonomy support. The study partner subscale is reported.
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale
  Baseline | 3.62 (1.94)
  12 weeks | 6.05 (0.94)

11. Secondary Outcome: Physical Activity Related Autonomy Support as Assessed by the Climate Questionnaire (Autonomy Support - Self Support Subscale)
Description: The Climate questionnaire (autonomy support) asses the level of autonomy support provided by both the individual (self) and their study partner. All participants completed both subscales: self-support and study partner support. The self support subscale is a 6 item questionnaire and each is scored from 1 (strongly disagree) to 7 (strongly agree). The sum of the 6 items were divided by 6, to generate a scale from 1 to 7, with higher scores indicating greater autonomy support. The self support subscale reported.
Time Frame: Baseline, 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale
  Baseline | 3.88 (1.97)
  12 weeks | 5.99 (0.89)

12. Secondary Outcome: Cognitive Impairment as Measured by the Montreal Cognitive Assessment (MoCA)
Description: Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Time Frame: 12 weeks
Population: Includes all twenty individuals enrolled (participants and their study partners).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching
Number analyzed (Participants) | 20
score on a scale | 25.9 (2.74)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Health Coaching
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05966506/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT05966506/ICF_001.pdf